CLINICAL TRIAL: NCT03940586
Title: A Phase 2b Open-label, Single-arm Study to Evaluate Pharmacokinetics, Efficacy, Safety and Tolerability of Letermovir in Pediatric Participants From Birth to Less Than 18 Years of Age at Risk of Developing CMV Infection and/or Disease Following Allogeneic Haematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Letermovir Treatment in Pediatric Participants Following Allogeneic Haematopoietic Stem Cell Transplantation (HSCT) (MK-8228-030)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8228-030; MK-8228-030 (Other: Merck Protocol Number); 205242 (Registry Identifier: JAPIC-CTI); 2018-001326-25 (EudraCT Number)
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Cytomegalovirus (CMV) Infection
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Letermovir (Experimental): Letermovir administered either orally or intravenously within 28 days post-transplant, once daily through week 14 (approximately 100 days). Dosing will vary based on age, weight, and whether participant takes cyclosporin A as a concomitant medication.
  Interventions: Drug: Letermovir oral granules; Drug: Letermovir tablet; Drug: Letermovir intravenous

INTERVENTIONS:
Drug: Letermovir oral granules — Granules administered orally based on age, weight, and whether participant takes cyclosporin A as a concomitant medication.
  Other Names: MK-8228; AIC246; AIC001
Drug: Letermovir tablet — Tablet administered orally based on age, weight, and whether participant takes cyclosporin A as a concomitant medication.
  Other Names: MK-8228; AIC246; AIC001
Drug: Letermovir intravenous — Letermovir administered intravenously based on age, weight, and whether participant takes cyclosporin A as a concomitant medication.
  Other Names: MK-8228; AIC246; AIC001

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) of letermovir (LET) in pediatric participants. Participants will be enrolled in the following 3 age groups: Age Group 1: From 12 to <18 years of age (adolescents); Age Group 2: From 2 to <12 years of age (children); and Age Group 3: From birth to <2 years of age (neonates, infants and toddlers). All participants will receive open label LET for 14 weeks (~100 days) post-transplant, with doses based on body weight and age.

ELIGIBILITY:
Inclusion Criteria:

* All participants 12 to <18 years old must have documented positive CMV serostatus (CMV IgG seropositive) for the recipient (R+) within 90 days prior to enrollment. Participants from birth to <12 years old must have documented positive CMV serostatus (CMV IgG seropositive) for the recipient (R+) within 90 days prior to enrollment and/or the donor (D+); the donor serostatus should be documented within 1 year prior to enrollment.
* Is the recipient of a first allogeneic HSCT (bone marrow, peripheral blood stem cell, or cord blood transplant).
* Has undetectable CMV DNA from a plasma or whole blood sample collected within 5 days prior to enrollment.
* Is within 28 days post-HSCT at the time of enrollment.
* Females are not pregnant, not breastfeeding,and is not a woman of childbearing potential (WOCBP); or is a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 28 days after the last dose of study intervention.
* Participants from 2 to <18 years of age must not be on concomitant Cyclosporin A (CsA), and must be able to take LET tablets or the oral granules (either by mouth or via G tube/NG tube), provided the participant does not have a condition that may interfere with the absorption of oral medication (e.g. vomiting, diarrhea, or a malabsorptive condition) from the day of enrollment until the intensive PK sampling is completed in these participants.
* For participants 2 <12 years old their weight should be at least 10 kg; for participants from birth to <2 years old their weight should be at least 2.5 kg and less than or equal to 15 kg at the time of enrollment.

Exclusion Criteria:

* Has received a previous allogeneic HSCT (Note: receipt of a previous autologous HSCT is acceptable).
* Has a history of CMV end-organ disease within 6 months prior to enrollment.
* Has evidence of CMV viremia at any time from either signing of the ICF or the HSCT procedure, whichever is earlier, until the time of enrollment.
* Has suspected or known hypersensitivity to active or inactive ingredients of LET formulations.
* Has severe hepatic insufficiency within 5 days prior to enrollment.
* Is a) on renal replacement therapy (eg, hemodialysis, peritoneal dialysis) OR b) has end-stage renal impairment.
* Has both moderate hepatic insufficiency and moderate-to-severe renal insufficiency.
* Has an uncontrolled infection on the day of enrollment.
* Requires mechanical ventilation or is hemodynamically unstable at the time of enrollment.
* Has a documented positive result for a human immunodeficiency virus antibody (HIVAb) test at any time prior to enrollment, or for hepatitis C virus antibody (HCV-Ab) with detectable HCV RNA, or hepatitis B surface antigen (HBsAg) within 90 days prior to enrollment.
* Has active solid tumor malignancies with the exception of localized basal cell or squamous cell skin cancer or the condition under treatment (e.g. lymphomas).
* Has a preexisting cardiac condition a) for which the patient is currently being treated or b) which required hospitalization within the last 6 months or c) that may be expected to recur during the course of the trial.
* Has received within 7 days prior to screening any of the following: ganciclovir; valganciclovir; foscarnet; acyclovir; valacyclovir; famciclovir.
* Has received within 30 days prior to screening of any of the following: cidofovir; CMV immunoglobulin; any investigational CMV antiviral agent/biologic therapy; Rifampin and other strong inducers (such as phenytoin, carbamazepine, St John's wort (Hypericum perforatum), rifabutin and phenobarbital) and moderate inducers such as nafcillin, thioridazine, modafinil and bosentan.
* Has received LET at any time prior to enrollment in this study.
* Is currently participating or has participated in a study with an unapproved investigational compound or device within 28 days, or 5X half-life of the investigational compound (excluding monoclonal antibodies), whichever is longer, of initial dosing in this study.
* Has previously participated in this study or any other study involving LET.
* Has previously participated or is currently participating in any study involving administration of a CMV vaccine or another CMV investigational agent, or is planning to participate in a study of a CMV vaccine or another CMV investigational agent during the course of this study.
* Is pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through 28 days after the last dose of study intervention.
* Is expecting to donate eggs starting from the time of consent through 28 days after the last dose of study intervention.
* Has clinically relevant drug or alcohol abuse within 12 months of screening that may interfere with participant treatment, assessment, or compliance with the protocol, as assessed by the investigator.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (40):
- United States (11):
  - City of Hope Comprehensive Cancer Center ( Site 0251), Duarte, California
  - Children's Hospital of Orange County ( Site 0241), Orange, California
  - UCSF Benioff Children's Hospital San Francisco ( Site 0245), San Francisco, California
  - University Of Chicago School Of Medicine ( Site 0253), Chicago, Illinois
  - Boston Children's Hospital ( Site 0243), Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center ( Site 0254), New York, New York
  - Duke University Health System ( Site 0252), Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center ( Site 0244), Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC ( Site 0258), Pittsburgh, Pennsylvania
  - Children's Medical Center ( Site 0257), Dallas, Texas
  - Seattle Childrens Hospital ( Site 0248), Seattle, Washington
- Australia (3):
  - The Children s Hospital at Westmead ( Site 0185), Westmead, New South Wales
  - Lady Cilento Children s Hospital ( Site 0182), South Brisbane, Queensland
  - Royal Childrens Hospital Melbourne ( Site 0181), Parkville, Victoria
- Colombia (3):
  - Instituto De Cancerologia S.A. ( Site 0213), Medellín, Antioquia
  - Fundacion Valle del Lili ( Site 0212), Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A ( Site 0211), Cali, Valle del Cauca Department
- Hôpital Universitaire Necker Enfants Malades-, Unite d'Immunologie-Hematologie et Rhumatologie Pedi, Paris, France
- Germany (4):
  - Universitaetsklinikum Frankfurt ( Site 0112), Frankfurt am Main, Hesse
  - Universitaetsklinikum Muenster ( Site 0114), Münster, North Rhine-Westphalia
  - Charite Universitaetsmedizin Berlin - Campus-Virchow-Klinikum ( Site 0113), Berlin
  - Universitatsklinikum Hamburg-Eppendorf ( Site 0111), Hamburg
- Israel (3):
  - Rambam Medical Center ( Site 0121), Haifa
  - Schneider Children's Medical Center ( Site 0122), Petah Tikva
  - Pediatric Hemato Oncology Safra Children's Hospital, Sheba Medical Center ( Site 0123), Ramat Gan
- Japan (2):
  - Saitama Children's Medical Center ( Site 0202), Saitama
  - National Center for Child Health and Development ( Site 0201), Tokyo
- Mexico (4):
  - Nuevo Hospital Civil Dr Juan I Menchaca ( Site 0223), Guadalajara, Jalisco
  - Instituto Nacional de Pediatria ( Site 0224), Mexico City, Mexico City
  - Hospital Infantil de Mexico ( Site 0221), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" ( Site 0222), Monterrey, Nuevo León
- Poland (2):
  - Szpital Uniwersytecki nr 1 im. Dr. Antoniego Jurasza w Bydgoszczy ( Site 0141), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckieg-Klinika Transplantacji Szpiku, Onkolog, Wroclaw, Lower Silesian Voivodeship
- Spain (4):
  - H. de la Santa Creu I Sant Pau ( Site 0155), Barcelona
  - Hospital Universitari Vall d Hebron ( Site 0154), Barcelona
  - Hospital Infantil Universitario Nino Jesus ( Site 0151), Madrid
  - Hospital Universitario La Paz ( Site 0153), Madrid
- Turkey (Türkiye) (3):
  - Acibadem Adana Hastanesi ( Site 0162), Adana
  - Akdeniz University Faculty of Medicine ( Site 0161), Antalya
  - Ege Univ.Tip Fakultesi Cocuk Has ( Site 0163), Izmir

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Groll AH, Schulte JH, Antmen AB, Fraser CJ, Teal VL, Haber B, Caro L, McCrea JB, Fancourt C, Patel M, Menzel K, Badshah C. Pharmacokinetics, Safety, and Efficacy of Letermovir for Cytomegalovirus Prophylaxis in Adolescent Hematopoietic Cell Transplantation Recipients. Pediatr Infect Dis J. 2024 Mar 1;43(3):203-208. doi: 10.1097/INF.0000000000004208. Epub 2024 Jan 19. PMID 38241643
- [Derived] Groll AH, Danziger-Isakov L, Gefen A, Fraser CJ, Schulte JH, Bielorai B, Karras NA, Bueno D, Shaw PJ, Broyde N, Haber B, Gilbert CL, Patel M, McCrea JB, Badshah C. Cytomegalovirus prophylaxis with letermovir in pediatric (birth to <18 years of age) hematopoietic cell transplant recipients: pharmacokinetics, efficacy, and safety results of a Phase 2b study. Antimicrob Agents Chemother. 2025 Oct;69(10):e0042025. doi: 10.1128/aac.00420-25. Epub 2025 Aug 18. PMID 40824644
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female recipients of a first allogeneic hematopoietic stem cell transplant (HSCT), between the ages of birth and <18 years of age, who were at risk for cytomegalovirus (CMV) infection and/or disease, and who had undetectable CMV deoxyribonucleic acid (DNA) collected within 5 days before enrollment. were enrolled in this study.
Groups:
- 12 - <18 Years: Letermovir (LET) 480 mg without cyclosporin (CsA), or 240 mg with CsA, administered either orally as tablets or in granular form, or by intravenous (IV) infusion, once daily (QD) through week 14 (~ 100 days) post-transplant.
- 2 - <12 Years: Participants ≥30 kg body weight (BW): LET 480 mg orally without CsA, or 240 mg with CsA, in granular form, or 240 mg IV with or without CsA; 18 to <30 kg BW: LET 240 mg orally without CsA, or 120 mg with CsA, either in granular form, or 120 mg IV with or without CsA; 10 to <18 kg BW: LET 120 mg orally without CsA, or 60 mg with CsA, in granular form, or 60 mg IV with or without CsA, all QD through week 14 (~ 100 days) post-transplant.
- Birth - <2 Years: 10 to ≤15 kg BW: LET 120 mg orally without CsA, or 60 mg with CsA, in granular form, or 60 mg IV with or without CsA; 7.5 to <10 kg BW: LET 80 mg orally without CsA, or 40 mg with CsA, either in granular form, or 40 mg IV with or without CsA; 5.0 to <7.5 kg BW: LET 40 mg orally without CsA, or 20 mg with CsA, in granular form, or 20 mg IV with or without CsA; 2.5 to <5.0 kg BW: LET 20 mg orally without CsA, or 10 mg with CsA, in granular form, or 10 mg IV with or without CsA, all QD through week 14 (~ 100 days) post-transplant.
Period: Overall Study
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Started (Randomized) | 28 | 29 | 8
Treated | 28 | 27 | 8
Completed (Through Week 48) | 21 | 21 | 6
Not Completed | 7 | 8 | 2
Not completed — Death | 3 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal By Parent/Guardian | 3 | 4 | 1
Not completed — Not Treated | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Treated Participants
Groups:
- 12 - <18 Years: LET 480 mg without CsA, or 240 mg with CsA, administered either orally as tablets or in granular form, or by IV infusion, QD through week 14 (~ 100 days) post-transplant.
- 2 - <12 Years: Participants ≥30 kg BW: LET 480 mg orally without CsA, or 240 mg with CsA, in granular form, or 240 mg IV with or without CsA; 18 to <30 kg BW: LET 240 mg orally without CsA, or 120 mg with CsA, either in granular form, or 120 mg IV with or without CsA; 10 to <18 kg BW: LET 120 mg orally without CsA, or 60 mg with CsA, in granular form, or 60 mg IV with or without CsA, all QD through week 14 (~ 100 days) post-transplant.
- Total: Total of all reporting groups
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years | Total
Number analyzed (Participants) | 28 | 27 | 8 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.1 (1.5) | 6.6 (3.2) | 0.7 (0.3) | 9.1 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 1 | 19
  Male | 15 | 22 | 7 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 1 | 14
  Not Hispanic or Latino | 14 | 21 | 6 | 41
  Unknown or Not Reported | 5 | 2 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 3 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 15 | 22 | 7 | 44
  More than one race | 4 | 2 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours Post-dose (AUC0-24) of Plasma Letermovir Taken as Oral Formulation by Ages 2 - <18 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 - <18 years in order to determine the AUC0-24 of plasma letermovir for participants receiving oral formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged < 2 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: All participants with at least one measurable PK sample who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements and absence of important protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- 12 - <18 Years: LET 480 mg without CsA as tablets or in granular form, was administered orally, QD through week 14 (~ 100 days) post-transplant.
- 2 - <12 Years: Participants 18 to <30 kg BW)received LET 240 mg without CsA orally in granular form QD through week 14 (~ 100 days) post-transplant.
- Birth - <2 Years: Participants 5 to <7.5 kg BW received LET 60 mg orally without CsA, in granular form, QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 5 | 4 | 0
hr*ng/mL | 80300 (74.9) | 62900 (37.4) |

2. Primary Outcome: AUC0-24 of Plasma Letermovir Taken as Oral Formulation by Ages 2 to <12 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 to <12 years in order to determine the AUC0-24 of plasma letermovir for participants receiving oral formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged <2 and >12 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: hr*ng/mL
Groups:
- 12 - <18 Years: LET 480 mg without CsA in tablet or granular form, was administered orally, QD through week 14 (~ 100 days) post-transplant.
- 2 - <12 Years: Participants 10 to <18 kg BW received LET 120 mg without CsA orally in granular form QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 2 | 0
hr*ng/mL |  | 39500 [23900 to 65200] |

3. Primary Outcome: AUC0-24 of Plasma Letermovir Taken as Oral Formulation by Ages <2 Years
Description: Blood was collected on treatment Day 7 from participants aged <2 years in order to determine the AUC0-24 of plasma letermovir for participants receiving oral formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged 2 - <18 years were not presented as their data analysis resulted in a different measure type and method of dispersion. The measure of dispersion is not determined when N <2.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: hr*ng/mL
Groups:
- 2 - <12 Years: Participants 18 to <30 kg BW received LET 240 mg without CsA orally in granular form QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 0 | 1
hr*ng/mL |  |  | 26200

4. Primary Outcome: Maximal Concentration (Cmax) of Plasma Letermovir Taken as Oral Formulation by Ages 2 - <18 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 - <18 years in order to determine the Cmax of plasma letermovir for participants receiving oral formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged < 2 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Birth - <2 Years: Participants 7.5 to <10 kg BW received LET 40 mg orally without CsA, in granular form, QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 5 | 4 | 0
ng/mL | 7410 (70.1) | 10800 (17.4) |

5. Primary Outcome: Cmax of Plasma Letermovir Taken as Oral Formulation by Ages 2 to <12 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 to <12 years in order to determine Cmax of plasma letermovir for participants receiving oral formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged <2 and >12 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 2 | 0
ng/mL |  | 5500 [5430 to 5580] |

6. Primary Outcome: Cmax of Plasma Letermovir Taken as Oral Formulation by Ages < 2 Years
Description: Blood was collected on treatment Day 7 from participants aged <2 years in order to determine the Cmax of plasma letermovir for participants receiving oral formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged 2 - <18 years were not presented as their data analysis resulted in a different measure type and method of dispersion. The measure of dispersion is not determined when N <2
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: ng/mL
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 0 | 1
ng/mL |  |  | 2950

7. Primary Outcome: Minimum Concentration of Plasma Letermovir Observed Before Next Dose (Ctrough) Taken as Oral Formulation by Ages 2 - <18 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 - <18 years in order to determine the Ctrough of plasma letermovir for participants receiving oral formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged < 2 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 5 | 4 | 0
ng/mL | 845 (107.5) | 171 (2046.8) |

8. Primary Outcome: Ctrough of Plasma Letermovir Taken as Oral Formulation by Ages 2 to <12 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 to <12 years in order to determine Ctrough of plasma letermovir for participants receiving oral formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged <2 and >12 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 2 | 0
ng/mL |  | 481 [207 to 1120] |

9. Primary Outcome: Ctrough of Plasma Letermovir Taken as Oral Formulation by Ages < 2 Years
Description: Blood was collected on treatment Day 7 from participants aged <2 years in order to determine the Ctrough of plasma letermovir for participants receiving oral formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged 2 - <18 years were not presented as their data analysis resulted in a different measure type and method of dispersion. The measure of dispersion is not determined when N <2.
Time Frame: Day 7: 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: ng/mL
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 0 | 1
ng/mL |  |  | 61.7

10. Primary Outcome: AUC0-24 of Plasma Letermovir Taken as Intravenous (IV) Formulation by Ages 12 - <18 Years
Description: Blood was collected on treatment Day 7 from participants aged 12 - <18 years in order to determine the AUC0-24 of plasma letermovir for participants receiving IV formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged < 12 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- 12 - <18 Years: LET 480 mg without CsA was administered by IV, QD through week 14 (~ 100 days) post-transplant.
- 2 - <12 Years: Participants 18 to <30 kg BW received LET 240 mg without CsA by IV QD through week 14 (~ 100 days) post-transplant.
- Birth - <2 Years: Participants 7.5 to <10 kg BW received LET 40 mg without CsA, by IV, QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 3 | 0 | 0
hr*ng/mL | 114000 (37.8) |  |

11. Primary Outcome: AUC0-24 of Plasma Letermovir Taken as IV Formulation by Ages 2 to <12 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 to <12 years in order to determine the AUC0-24 of plasma letermovir for participants receiving IV formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged < 2 years and > 12 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: hr*ng/mL
Groups:
- 2 - <12 Years, ≥30 kg BW: Participants ≥30 kg BW received LET 240 mg without CsA orally by IV QD through week 14 (~ 100 days) post-transplant.
- 2 - <12 Years, 18 to <30 kg BW: Participants 18 to <30 kg BW received LET 120 mg without CsA, by IV QD through week 14 (~ 100 days) post-transplant.
- Birth - <2 Years: Participants 5.0 to <7.5 kg BW received LET 40 mg without CsA, by IV QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years, ≥30 kg BW | 2 - <12 Years, 18 to <30 kg BW | Birth - <2 Years
Number analyzed (Participants) | 0 | 2 | 2 | 0
hr*ng/mL |  | 36200 [21000 to 62100] | 31500 [20300 to 48900] |

12. Primary Outcome: AUC0-24 of Plasma Letermovir Taken as IV Formulation by Ages 2 to <12 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 to <12 years in order to determine the AUC0-24 of plasma letermovir for participants receiving IV formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged > 2 years were not presented as their data analysis resulted in a different measure type and method of dispersion. The measure of dispersion is not determined when N <2.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: hr*ng/mL
Groups:
- 2 - <12 Years: Participants 10 to <18 kg BW received LET 60 mg without CsA by IV QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 1 | 0
hr*ng/mL |  | 25300 |

13. Primary Outcome: AUC0-24 of Plasma Letermovir Taken as IV Formulation by Ages <2 Years
Description: Blood was collected on treatment Day 7 from participants aged <2 years in order to determine the AUC0-24 of plasma letermovir for participants receiving IV formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged > 2 years were not presented as their data analysis resulted in a different measure type and method of dispersion. The measure of dispersion is not determined when N <2.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: hr*ng/mL
Groups:
- 2 - <12 Years: Participants ≥30 kg BW received LET 240 mg without CsA by IV QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 0 | 1
hr*ng/mL |  |  | 37300

14. Primary Outcome: Concentration at the End of Infusion (Ceoi) of Plasma Letermovir Taken as IV Formulation by Ages 12 - <18 Years
Description: Blood was collected on treatment Day 7 from participants aged 12 - <18 years in order to determine the Ceoi of plasma letermovir for participants receiving IV formulation. As samples were collected outside the collection window Ceoi for these samples were predicted by using a log linear model .Participants aged < 12 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Birth - <2 Years: Participants 7.5 to <10 kg BW received LET 40 mg orally without CsA, by IV, QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 3 | 0 | 0
ng/mL | 30600 (16.4) |  |

15. Primary Outcome: Ceoi of Plasma Letermovir Taken as IV Formulation by Ages 2 to <12 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 to <12 years in order to determine the Ceoi of plasma letermovir for participants receiving IV formulation. As samples were collected outside the collection window Ceoi for these samples were predicted by using a log linear model. Participants aged < 2 years and > 12 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- 2 - <12 Years, 18 to <30 kg BW: Participants18 to <30 kg BW received LET 120 mg without CsA by IV QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years, ≥30 kg BW | 2 - <12 Years, 18 to <30 kg BW | Birth - <2 Years
Number analyzed (Participants) | 0 | 2 | 2 | 0
ng/mL |  | 16800 [14900 to 19000] | 8200 [7580 to 8870] |

16. Primary Outcome: Ceoi of Plasma Letermovir Taken as IV Formulation by Ages s 2 to <12 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 to <12 years in order to determine the Ceoi of plasma letermovir for participants receiving IV formulation. As samples were collected outside the collection window Ceoi for these samples were predicted by using a log linear model. Participants aged > 2 years were not presented as their data analysis resulted in a different measure type and method of dispersion. A measure of dispersion is not determined when N <2.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: ng/mL
Groups:
- 2 - <12 Years: Participants 10 to < 18 kg body BW received LET 60 mg without CsA by IV QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 1 | 0
ng/mL |  | 8630 |

17. Primary Outcome: Ceoi of Plasma Letermovir Taken as IV Formulation by Ages <2 Years
Description: Blood was collected on treatment Day 7 from participants aged <2 years in order to determine the Ceoi of plasma letermovir for participants receiving IV formulation. As samples were collected outside the collection window Ceoi for these samples were predicted by using a log linear model. Participants aged > 2 years were not presented as their data analysis resulted in a different measure type and method of dispersion. A measure of dispersion is not determined when N <2.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: ng/mL
Groups:
- 2 - <12 Years: Participants ≥30 kg body BW received LET 240 mg without CsA by IV QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 0 | 1
ng/mL |  |  | 11700

18. Primary Outcome: Ctrough of Plasma Letermovir Taken as IV Formulation by Ages 12 - <18 Years
Description: Blood was collected on treatment Day 7 from participants aged 12 - <18 years in order to determine the Ctrough of plasma letermovir for participants receiving IV formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged < 12 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 3 | 0 | 0
ng/mL | 709 (256.8) |  |

19. Primary Outcome: Ctrough of Plasma Letermovir Taken as IV Formulation by Ages 2 to <12 Years
Description: Blood was collected on treatment Day 7 from participants aged 2 to <12 years in order to determine the Ctrough of plasma letermovir for participants receiving IV formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged < 2 years and > 12 years were not presented as their data analysis resulted in a different measure type and method of dispersion.
Time Frame: Day 7: 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- 2 - <12 Years, ≥30 kg BW: Participants ≥30 kg BW received LET 240 mg without CsA by IV QD through week 14 (~ 100 days) post-transplant.
- 2 - <12 Years,18 to <30 kg BW: Participants 18 to <30 kg BW received LET 120 mg without CsA by IV QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years, ≥30 kg BW | 2 - <12 Years,18 to <30 kg BW | Birth - <2 Years
Number analyzed (Participants) | 0 | 2 | 2 | 0
ng/mL |  | 71.6 [12.9 to 397] | 318 [134 to 754] |

20. Primary Outcome: Ctrough of Plasma Letermovir Taken as IV Formulation by Ages 2 to <12 Years
Description: Blood was collected on treatment Day 7 from participants aged <2 years in order to determine the Ctrough of plasma letermovir for participants receiving IV formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged > 2 years were not presented as their data analysis resulted in a different measure type and method of dispersion. The measure of dispersion is not determined when N <2.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: ng/mL
Groups:
- 2 - <12 Years: Participants 10 to < 18 kg BW received LET 60 mg without CsA by IV QD through week 14 (~ 100 days) post-transplant.
- Birth - <2 Years: Participants 5.0 to <7.5 kg BW received LET 40 mg with CsA, by IV QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 1 | 0
ng/mL |  | 216 |

21. Primary Outcome: Ctrough of Plasma Letermovir Taken as IV Formulation by Ages <2 Years
Description: Blood was collected on treatment Day 7 from participants aged <2 years in order to determine the Ctrough of plasma letermovir for participants receiving IV formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant. Participants aged > 2 years were not presented as their data analysis resulted in a different measure type and method of dispersion. The measure type is Geometric Mean, and a measure of dispersion is not determined when N <2.
Time Frame: Day 7: Pre-dose, 1, 2.5, 8, and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: ng/mL
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 0 | 1
ng/mL |  |  | 98.3

22. Primary Outcome: Ctrough of Plasma Letermovir Taken During Sparse PK for Oral Formulation
Description: Blood was collected on treatment Day 7 in order to determine the Ctrough of plasma letermovir during sparse PK for participants receiving oral formulation. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant.
Time Frame: Day 7: 24 hours post-dose
Population: Per protocol, sparse PK results were not planned as either primary or secondary outcome measures. As sparse PK data were instead used in population PK model development, they were not summarized in this outcome measure.
Groups:
- 12 - <18 Years: LET 480 mg administered orally by tablet or granular form within 28 days post-transplant, QD with or without CsA through week 14 (approximately 100 days).
- 2 - <12 Years; Birth - <2 Years: LET administered orally in granular form without CsA within 28 days post-transplant, QD through week 14 (approximately 100 days). Dosing varied based on weight.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 0 | 0

23. Primary Outcome: Ctrough of Plasma Letermovir Taken During Sparse PK as IV Formulation
Description: Blood was collected on treatment Day 7 in order to determine the Ctrough of plasma letermovir for participants receiving IV formulation during sparse PK. Individual values were natural log transformed and evaluated separately with a linear mixed effects model containing a fixed effect for treatment and a random effect for participant.
Time Frame: Day 7: 24 hours post-dose
Population: as for outcome 22
Groups:
- 12 - <18 Years: LET 480 mg administered by IV within 28 days post-transplant, QD without CsA through week 14 (approximately 100 days).
- 2 - <12 Years: LET administered by IV within 28 days post-transplant, QD without CsA through week 14 (approximately 100 days). Dosing varied based on weight.
- Birth - <2 Years: LET administered by IV without CsA within 28 days post-transplant, QD through week 14 (approximately 100 days). Dosing varied based on weight.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Percentage of Participants With One or More Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The 95% confidence interval (CI) is based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to Week 48 post-transplant (up to 52 weeks)
Population: All participants who received ≥1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 12 - <18 Years: LET 480 mg without CsA, or 240 mg with CsA, administered either orally in tablet or granular form, or by IV infusion, QD through week 14 (~ 100 days) post-transplant.
- 2 - <12 Years: ≥30 kg body BW: LET 480 mg orally without CsA, or 240 mg with CsA, in granular form, or 240 mg IV with or without CsA; 18 to <30 kg BW: LET 240 mg orally without CsA, or 120 mg with CsA, either in granular form, or 120 mg IV with or without CsA; 10 to <18 kg BW: LET 120 mg orally without CsA, or 60 mg with CsA, in granular form, or 60 mg IV with or without CsA, all QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 28 | 27 | 8
Percentage of participants | 100.0 [87.7 to 100.0] | 100.0 [87.7 to 100.0] | 100.0 [63.1 to 100.0]

25. Secondary Outcome: Percentage of Participants Who Discontinued Study Medication Due to an AE.
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The 95% CI is based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to Week 14 post-transplant (up to 18 weeks)
Population: All participants who received ≥1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 2 - <12 Years: ≥30 kg BW: LET 480 mg orally without CsA, or 240 mg with CsA, in granular form, or 240 mg IV with or without CsA; 18 to <30 kg BW: LET 240 mg orally without CsA, or 120 mg with CsA, either in granular form, or 120 mg IV with or without CsA; 10 to <18 kg BW: LET 120 mg orally without CsA, or 60 mg with CsA, in granular form, or 60 mg IV with or without CsA, all QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 28 | 27 | 8
Percentage of participants | 17.9 [6.1 to 36.9] | 7.4 [0.9 to 24.3] | 12.5 [0.3 to 52.7]

26. Secondary Outcome: Percentage of Participants With Clinically Significant CMV Infection Through Week 14 Post-transplant
Description: Clinically significant cytomegalovirus (CMV) infection is defined as CMV end organ disease (proven or probable) or initiation of pre-emptive therapy (PET) based on documented CMV viremia and the clinical condition of the participant. The 95% confidence interval (CI) was based on the exact binomial method proposed by Clopper and Pearson. Missing values: were handled by the Non-Completer=Failure (NC=F) approach. where failure was defined as all participants who developed clinically significant CMV infection or prematurely discontinued from the study or had a missing outcome through week 14 post-transplant visit window.
Time Frame: Up to Week 14 post-transplant (up to 18 weeks)
Population: Participants who received ≥1 dose of study intervention, had no detectable CMV viral DNA on the day study intervention was initiated, had not prematurely discontinued from the study and had an outcome through week 14 post-transplant.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 25 | 24 | 7
Percentage of participants | 20.0 [6.8 to 40.7] | 16.7 [4.7 to 37.4] | 28.5 [3.7 to 71.0]

27. Secondary Outcome: Percentage of Participants With Clinically Significant CMV Infection Through Week 24 Post-transplant
Description: Clinically significant CMV infection is defined as CMV end organ disease (proven or probable) or initiation of PET based on documented CMV viremia and the clinical condition of the participant. The 95% confidence interval (CI) was based on the exact binomial method proposed by Clopper and Pearson. Missing values: were handled by the Non-Completer=Failure (NC=F) approach. where failure was defined as all participants who developed clinically significant CMV infection or prematurely discontinued from the study or had a missing outcome through week 24 post-transplant visit window.
Time Frame: Up to Week 24 post-transplant (up to 28 weeks)
Population: Participants who received ≥1 dose of study intervention, had no detectable CMV viral DNA on the day study intervention was initiated, had not prematurely discontinued from the study and had an outcome through week 24 post-transplant.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 12 - <18 Years: LET 480 mg without CsA, or 240 mg with CsA, administered either orally in tablet or granular form, or IV infusion, QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 25 | 24 | 7
Percentage of participants | 24.0 [9.4 to 45.1] | 25.0 [9.8 to 46.7] | 28.6 [3.7 to 71.0]

28. Secondary Outcome: Number of Participants Receiving Oral Granules With Palatability Response, Based on Taste of Medication on the First Day of Administration of Oral Formulation
Description: Palatability was measured by response to a questionnaire on the taste of medication , with responses from very good, good, neither good nor bad, bad or very bad.
Time Frame: Day 1 of administration of oral formulation up to Week 14 post-transplant (up to 18 weeks)
Population: Participants who received ≥1 dose of study intervention, and completed palatability questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 4 | 27 | 7
Participants
  Very good | 0 | 3 | 0
  Good | 1 | 5 | 3
  Neither good nor bad | 1 | 8 | 1
  Bad | 1 | 8 | 3
  Very bad | 1 | 3 | 0

29. Secondary Outcome: Number of Participants Receiving Oral Granules With Palatability Response, Based on Taste of Medication on the Eighth Day of Administration of Oral Formulation
Description: as for outcome 28
Time Frame: Day 8 of administration of oral formulation up to Week 14 post-transplant (up to 18 weeks)
Population: Participants who received ≥1 dose of study intervention, and completed palatability questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | 12 - <18 Years | 2 - <12 Years | Birth - <2 Years
Number analyzed (Participants) | 2 | 23 | 7
Participants
  Very good | 0 | 3 | 0
  Good | 1 | 4 | 3
  Neither good nor bad | 1 | 8 | 4
  Bad | 0 | 5 | 0
  Very bad | 0 | 3 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM): from allocation/randomization (i.e. prior to treatment) up to Week 48 post-transplant (up to 52 weeks). AEs: From first treatment up to Week 48 post-transplant (up to 52 weeks)
Description: ACMs: the population analyzed was all allocated/randomized participants. AEs: the population analyzed was all allocated/randomized participants who received ≥1 dose of study intervention.
Groups:
- <2 Years: 10 to ≤15 kg BW: LET 120 mg orally without CsA, or 60 mg with CsA, in granular form, or 60 mg IV with or without CsA; 7.5 to <10 kg BW: LET 80 mg orally without CsA, or 40 mg with CsA, either in granular form, or 40 mg IV with or without CsA; 5.0 to <7.5 kg BW: LET 40 mg orally without CsA, or 20 mg with CsA, in granular form, or 20 mg IV with or without CsA; 2.5 to <5.0 kg BW: LET 20 mg orally without CsA, or 10 mg with CsA, in granular form, or 10 mg IV with or without CsA, all QD through week 14 (~ 100 days) post-transplant.
Arm/Group | 12 - <18 Years | 2 - <12 Years | <2 Years
All-Cause Mortality (participants affected / at risk) | 4/28 | 2/29 | 0/8
Serious Adverse Events (participants affected / at risk) | 13/28 | 18/27 | 7/8
Other Adverse Events (participants affected / at risk) | 27/28 | 27/27 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 - <18 Years (N=28) | 2 - <12 Years (N=27) | <2 Years (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 2 (2) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1) | 1 (2) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
BK virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatosplenic candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Human herpesvirus 6 infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Engraft failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Venoocclusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 - <18 Years (N=28) | 2 - <12 Years (N=27) | <2 Years (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 (5) | 8 (18) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (4) | 3 (6) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 9 (12) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (8) | 11 (11) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 3 (4) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (14) | 7 (11) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (7) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 14 (20) | 13 (20) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (25) | 8 (9) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 9 (9) | 9 (9) | 0 (0)
Vomiting (Gastrointestinal disorders) | 17 (47) | 21 (55) | 4 (6)
Asthenia (General disorders) | 1 (3) | 4 (7) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0)
Face oedema (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (3) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 11 (18) | 13 (25) | 4 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 3 (3) | 0 (0)
Engraftment syndrome (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Graft versus host disease (Immune system disorders) | 10 (14) | 10 (13) | 3 (3)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 0 (0) | 1 (2)
Adenovirus infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
BK virus infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Epstein-Barr virus infection reactivation (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Polyomavirus viraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 2 (3) | 2 (3) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (6) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 1 (1) | 1 (1)
BK polyomavirus test positive (Investigations) | 2 (2) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Cytomegalovirus test positive (Investigations) | 2 (2) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Immunosuppressant drug level increased (Investigations) | 0 (0) | 2 (7) | 0 (0)
Oxygen saturation decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (3) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (5) | 8 (10) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (7) | 5 (8) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (6) | 4 (5) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (7) | 4 (5) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (4) | 2 (3) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Neonatal diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Sodium retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (11) | 4 (5) | 0 (0)
Tremor (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (4) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 6 (6) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 2 (2) | 0 (0)
Hypercalciuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 3 (3) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (6) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (6) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail pigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (6) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 8 (10) | 10 (14) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 2 (3) | 0 (0)
Eye irritation (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (5) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT03940586/Prot_SAP_000.pdf